CLINICAL TRIAL: NCT06534801
Title: Sequential Method Determination of Oxycodone for Thoracoscope Surgery Median Effective Dose of Acute Pain Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianbo Wu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Wu, Chief Physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YXLL-KY-2024(058)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Oxycodone; Thoracoscopic Lobectomy; Acute Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I（Age < 65 years old) (Experimental): We will use the sequential allocation designed by Dixon. Oxycodone will be administered intravenously 30min before the end of surgery. The initial oxycodone dose will be set to 0.1 mg/kg. A satisfactory or an unsatisfactory analgesic response of the previous patient determined, respectively, the relative 10% decrease or increase in the dose of oxycodone the next patient received in the same group. The patient before the first crossover point will be included as the first case for ED50 estimation in each group. The study will conducted until 7 crossover points have be collected .
  Interventions: Drug: Oxycodone will be administered intravenously in the group 1
- Group II(Age ≥65 years old) (Experimental): We will use the sequential allocation designed by Dixon. Oxycodone will be administered intravenously 30min before the end of surgery. The initial oxycodone dose will be set to 0.1 mg/kg. A satisfactory or an unsatisfactory analgesic response of the previous patient determined, respectively, the relative 10% decrease or increase in the dose of oxycodone the next patient received in the same group. The patient before the first crossover point will be included as the first case for ED50 estimation in each group. The study will conducted until 7 crossover points have be collected .
  Interventions: Drug: Oxycodone will be administered intravenously in the group 1

INTERVENTIONS:
Drug: Oxycodone will be administered intravenously in the group 1 — Oxycodone will be administered intravenously 30min before the end of surgery, and Dixon sequential method will be used for the study
  Other Names: They are grouped according to age

SUMMARY:
The goal of this clinical trial is to measure the median effective dose of oxycodone for the treatment of acute pain after thoracoscopic lobectomy. This clinical trial was divided into two groups based on age, Group I (Age < 65 years old) and Group II (Age ≥65 years old). We used the sequential allocation designed by Dixon. The initial oxycodone dose was set to 0.1 mg/kg.A satisfactory or an unsatisfactory analgesic response of the previous patient determined, respectively, the relative 10% decrease or increase in the dose of oxycodone the next patient received in the same group. The patient before the first crossover point was included as the first case for ED50 estimation in each group.The study was conducted until 7 crossover points were collected

ELIGIBILITY:
Inclusion Criteria:

1. The first unilateral thoracoscopic lobectomy was performed under general anesthesia
2. age 18- 80 years old
3. American Society of Anesthesiologists (ASA) physical status I-III
4. Sign the informed consent of the patients

Exclusion Criteria:

1. Moderate to severe obesity (i.e., BMI > 30kg/m2)
2. Allergic or hypersensitive reaction to oxycodon
3. A history of chronic pain
4. Patients with significant heart, pulmonary, liver or renal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The median effective dose | 3 minutes after remoal of the endotracheal tube, 30minutes after remoal of the endotracheal tube
  The median effective dose of oxycodone for the treatment of acute pain after thoracoscopic lobectomy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Liu Y, Cao J, Liu M, Gao X, Guo N, Wei C, Zhu Y, Sun Y, Wu J. The median effective dose of oxycodone for acute postoperative pain after thoracoscopic pulmonary surgery with intercostal nerve blockin in patients of different ages: a dose-finding study protocol. BMC Anesthesiol. 2025 Jul 1;25(1):323. doi: 10.1186/s12871-025-03198-5. PMID 40597587